CLINICAL TRIAL: NCT07383012
Title: Long-term Follow-up Study to Evaluate the Long-term Safety and Performance of PCL Breast Scaffolds Used for Breast Implant Revision Surgery in 2021-BRV-004
Brief Title: LTFU of PCL Breast Scaffolds Used in 2021-BRV-004
Status: Not yet recruiting | Type: Observational
Sponsor: BellaSeno Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: BellaSeno GmbH (Industry)
Other Study IDs: 2025-BRV-006
Record Dates: First submitted 2026-01-15; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Breast Implant Revision
Keywords: Breast scaffold; PCL scaffold; Long-term Safety and Performance; Absorbable Implant; Regenerative Medicine; PCL breast scaffold; Mammography screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Core biopsies may be performed during the study if clinically indicated. De-identified biopsy samples will be collected and stored only after obtaining participant consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCL Breast Scaffold Follow-up Group: Participants from the 2021-BRV-004 study receiving long-term follow-up assessments at 3-, 4- and 5-years after implantation of the PCL Breast Scaffold

SUMMARY:
The objective of this study is to assess the long-term safety and performance of the PCL Breast Scaffold in women who previously underwent breast silicone implant revision and received the PCL Breast Scaffold combined with autologous fat grafting (AFG) in the 2021-BRV-004 clinical trial (ClinicalTrials.gov ID: NCT05437757). In addition, this study will investigate the suitability of mammography in the subset of patients that fall into the national breast screening age category - individuals aged 40 years and older.

The main questions this study aims to answer are:

* "Is the PCL Breast Scaffold combined with autologous fat grafting a safe and effective method of soft-tissue reconstruction following breast implant revision?"
* "Is mammography a suitable follow-up screening and diagnostic tool for patients implanted with the PCL Breast Scaffold?"

Participants will attend annual follow-up visits from 3 to 5 years after PCL Breast Scaffold implantation for clinical assessments and patient-reported outcome questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with at least one PCL Breast Scaffold who took part in the 2021-BRV-004 study.
* Patients who provide written informed consent to participate in this study.

Exclusion Criteria:

* Patient unwilling and unable to comply with the study requirements.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Study Population: Participants who took part in the 2021-BRV-004 study, meet the eligibility criteria and provide informed consent to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of moderate and severe device-related (probable and causal) AEs rate | Assessed at 3-, 4- and 5-years after implantation of the PCL Breast Scaffold
  Number of moderate and severe AEs with a probable or causal relationship to the device falling under pre-defined category over time

SECONDARY OUTCOMES:
Breast revision surgery rate | Assessed at 3-, 4- and 5-years after implantation of the PCL Breast Scaffold
  Number of breast revision surgeries categorized by reason and time
Rate and severity of all AEs related to device and/or procedure | Assessed at 3-, 4- and 5-years after implantation of the PCL Breast Scaffold
  Number of AEs categorised by relationship with device and/or procedure (possible, probable, causal), severity and type over time
Total breast volume retention (3D Imaging) | Assessed at 3- and 5-years after implantation of the PCL Breast Scaffold
  Total breast volume primarily assessed through 3D imaging. Supportive data generated by:
  * Dynamic contrast enhanced Magnetic Resonance Imaging (DCE-MRI)
  * Breast anthropomorphic measurements taken with tape measure or the Vectra imaging system (Sternal notch to nipple (SN-N), Nipple to inframammary fold (N-IMF), Overbust measurement, Underbust measurement, Chest circumference at highest projection)
  * Digital photos
Assessment of patient satisfaction, quality of life, body image, and psychological well-being using the validated BREAST-Q questionnaire | Assessed at 3-, 4- and 5-years after implantation of the PCL Breast Scaffold
  Patient-reported outcomes will be measured using the validated BREAST-Q questionnaire. Results are reported as a transformed score range from 0 to 100, with higher scores reflecting a better outcome.
Assessment of patient satisfaction, quality of life, body image, and psychological well-being using a 5-point Likert scale questionnaire | Assessed at 3-, 4- and 5-years after implantation of the PCL Breast Scaffold
  Patient-reported outcomes will be measured through a 5-point Likert scale questionnaire. Scores range from 1 to 5, with higher scores indicating better outcomes.
Assessment of device user experience using a 5-point Likert scale questionnaire | Assessed at 3-, 4- and 5-years after implantation of the PCL Breast Scaffold
  The 5-point Likert scale questionnaire is administered to the PI. Scores range from 1 to 5, with higher scores indicating greater surgeon satisfaction.
Assessment of suitability of mammography after scaffold implantation | Assessed at 3-, 4- and 5-years after implantation of the PCL Breast Scaffold
  Visibility of glandular breast tissue; visibility of all regions of interest required for effective screening; any interference caused by the scaffold that may affect the sensitivity and specificity of the diagnostic method; visibility of the scaffold or regenerated tissue; visibility of any findings previously detected by (DCE-)MRI; and visibility of any liquid formation or seroma, if present.

OTHER OUTCOMES:
Technical possibility of MRI for tracking scaffold degradation | Assessed at 3-, 4- and 5-years after implantation of the PCL Breast Scaffold
  Visibility of ongoing degradation compared to previous visit through DCE-MRI
Assessment of suitability of US (if medically indicated) screening after scaffold implantation | Only if medically indicated between 3 and 5 years after implantation of the PCL breast scaffold.
  Visibility of all regions of interest required for effective screening; any interference caused by the scaffold that affects the Color Doppler US reporting; visibility of the scaffold or regenerated tissue; visibility of any findings previously detected by DCE-MRI; and visibility of any liquid formation or seroma, including estimation of US-based calculated volume when present.
Biopsy, if clinically indicated, will be used for assessment of: tissue viability, tissue composition, tissue vascularisation, inflammatory response | Reccomended 3 years after implantation of the PCL Breast Scaffold
  Assessments include tissue viability (presence of viable cells and observation of any necrotic tissue), tissue composition (tissue type, presence of calcifications or oil cysts), tissue vascularization (presence of blood vessels), and inflammatory response (presence of inflammation and whether it is acute or chronic)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Owen Ung, Principal Investigator — Royal Brisbane and Women's Hospital (RBWH), Herston Biofabrication Institute (HBI)
Locations (1):
- Royal Brisbane and Women's Hospital (RBWH), Herston Biofabrication Institute (HBI), Brisbane, Queensland, Australia, Australia

IPD SHARING:
Plan to Share IPD: No